# Statistical Analysis Plan (SOP)

**Parent study Title:** "The Effect of Plasma Donation Frequency on Plasma Protein Composition, Inflammation Markers and Psychological Distress - a Randomized Controlled Trial"

**Sub Study Title:** "The Effect of Plasma Donation Frequency on PFAS Concentrations – a randomized controlled trial"

ClinicalTrials.gov Reference: NCT05179200

**Date:** 01.09.2025

### Introduction

# Background and Rationale

Poly- and perfluoroalkyl substances (PFAS) are synthetic compounds used for their water- and fat-repellent properties in products such as textiles, food packaging, cosmetics, and electronics [1-3]. PFAS are highly persistent in the environment and the human body, with long biological half-lives of 1-5 years [4]. As a result, they are widely detected in drinking water, soil, and food. Exposure in humans primarily occurs through the ingestion of contaminated water and food, as well as through everyday consumer products such as non-stick cookware, water-repellent clothing, food packaging, dental floss, and cosmetics. PFAS are absorbed into the bloodstream and bind to proteins rather than fat [3, 5-7], leading to bioaccumulation over time [1, 8]. This accumulation has been linked to adverse health effects, including immune suppression, hormonal disruption, elevated cholesterol, and potential carcinogenicity [9].

PFAS exposure is primarily assessed through blood concentrations. A recent Swedish study investigated PFAS exposure in the general population and analysed samples from 60 blood donors [10]. They detected 26 of 30 different PFAS and observed PFHxS-lin, PFOS (linear and branched), PFOA-lin, PFNA, and PFDA in all samples, and found the highest concentrations of PFOS-lin, PFOS-br, PFOA-lin, and PFHxS-lin.

A previous RCT in Australian firefighters, with high exposure to PFAS through firefighting foams, demonstrated reductions in PFAS concentrations following plasma donations every 6 weeks and blood donations every 12 weeks [11].

In this study, we aim to investigate the effect of different plasma donation frequencies on PFAS concentrations in blood donors.

# Objectives

To compare the plasma concentration of different PFAS at baseline and after 16 weeks of donations between high-frequency plasma donors (HFPDs), donating plasma 3 times every 2 weeks, regular-frequency plasma donors (RFPDs), donating plasma once every 2 weeks, and a control group (controls) donating whole blood every 3 months.

# Study Methods

## Trial Design

This is a randomized controlled trial, parallel-group, where 120 male blood donors were randomized 1:1:1 for donation over 16 weeks to:

- High-frequency plasma donors (HFPDs) donating plasma 3 times every 2 weeks (in total 24 times)
- Regular-frequency plasma donors (RFPDs) donating plasma once every 2 weeks (in total 8 times)
- The control group (controls) donating whole blood every 3 months (in total 2 times)

The study was conducted at the Blood Centre of Innlandet Hospital Trust from January 2022 to July 2024.

### **Trial Population**

Established male blood- and plasma donors aged between 18 and 64 years were screened for eligibility. The inclusion criteria were sufficient levels of Hb, TSP, and IgG, an estimated blood volume (EBV) of at least 4500 mL, a donation history of at least one previous plasma donation, and the donors had to meet the eligibility criteria for both whole blood and plasma donation by plasmapheresis. Donors with a history of repeated measurements (>2) of haematocrit >50 % before enrolment were excluded.

All participants provided written informed consent. The study was approved by the Regional Committee for Medical and Health Research Ethics in Southeast Norway (2021/238929/REC Southeast A) and was conducted in accordance with the Declaration of Helsinki. The study is registered at clinicaltrials.gov (identifier: NCT05179200).

#### Intervention

The plasmapheresis procedure was performed using the Aurora Plasmapheresis machine, Fresenius Kabi. The plasma donation volume was 720 mL, including AC, which corresponds to approximately 650 mL plasma, excluding AC, assuming a haematocrit of 44% and an ACR of 100:6. The whole blood donations were 450 mL of whole blood.

#### **Data Collection**

Baseline data were collected through questionnaires and from the blood centre's database, LabCraft.

#### **Blood Samples and Analyses**

One tube of 6 mL EDTA plasma was collected non-fasting per participant immediately before the plasmapheresis procedure, at:

- Baseline week 1 (W1): Before the first donation in the study, after at least two months of no donation.
- End point week 18 (W18): Two weeks after the final donation.

The plasma samples were centrifuged at  $2200 \times g$  for 10 min immediately after collection, transferred into aliquots of  $500~\mu\text{L}$ , and frozen at  $-40^{\circ}\text{C}$  within 3 hours after collection. Within 3 months of storage, the samples were transferred to storage at  $-80^{\circ}\text{C}$  until analysis. The samples were shipped on dry ice to the laboratory for analysis. PFAS analyses were conducted at the Environmental Pollutant Laboratory, University Hospital of North Norway, Tromsø, Norway, according to the method described by Huber and Brox [12]. Samples were analysed in two batches of 96 samples in 2023 and 122 samples in 2024.

### **Variables**

#### **Outcome Measures**

Difference in plasma concentrations between W1 and W18 of the following PFAS:

#### **Primary outcomes:**

- Perfluorooctanoic acid (PFOA)
- Perfluorooctane sulfonic acid (PFOS)\*
- Perfluorohexane sulfonic acid (PFHxS)\*
- Perfluorononanoic acid (PFNA)
- Sum of PFOA, PFOS, PFHxS and PFNA [13]

#### **Secondary outcomes:**

- Perfluorobutanoic acid (PFBA)
- Perfluoropentanoic acid (PFPeA)
- Perfluorohexanoic acid (PFHxA)
- Perfluoroheptanoic acid (PFHpA)
- Perfluorodecanoic acid (PFDA)
- Perfluoroundecanoic acid (PFUDA)
- Perfluorododecanoic acid (PFDoDA)
- Perfluorotridecanoic Acid (PFTrDA)
- Perfluorotetradecanoic acid (PFTeDA)
- Perfluorobutane sulfonic acid (PFBS)
- Perfluoropentane sulfonic acid (PFPS)
- Perfluorooctane sulfonic acid (PFHpS)\*
- Perfluorononane sulfonic acid (PFNS)\*
- Perfluorodecane sulfonic acid (PFDS)\*
- Perfluorodecane sulfonic acid (PFDoDS)
- Perfluorooctane sulfonamide (PFOSA)\*
- 4:2 Fluorotelomer sulfonic acid (4:2 FTSA)
- 6:2 Fluorotelomer sulfonic acid (6:2 FTSA)
- 8:2 Fluorotelomer sulfonic acid (8:2 FTSA )
- 10:2 Fluorotelomer sulfonic acid (10:2 FTSA)

#### Other variables:

• Plasma albumin concentration (as a mediator)

### Independent Variables

• Study group identity (HFPDs, RFPDs, control group)

<sup>\*</sup>Analysed as linear and branched isomers, and the sum of these.

# Statistical Analysis

Stata (StataCorp, College Station, TX, USA) will be used for the statistical analyses.

Outcome variables will be checked for normality. Normally distributed data will be expressed as mean (SD), and non-normally distributed data will be expressed as median (min-max and/or IQR). 95% confidence intervals will be used, and a two-tailed p-value < 0.05 will be considered statistically significant.

Samples below the detection and quantification limits:

- The number, n (%), of samples below the limit of quantification (LOQ), as defined per the laboratory protocol, will be calculated.
- The number, n (%), of samples below the limit of detection (LOD) will be calculated.
- Only PFAS (or summarized variables) with a detection rate >70% at baseline will be included in the statistical analysis [14, 15].

For values below the LOD, a common imputation approach will be used where concentrations are replaced by LOD/2 (i.e., one-half the detection limit). Sensitivity analyses may be conducted to evaluate the choice of imputation method for values below the LOD (e.g., LOD/2, LOD/ $\sqrt{2}$ , or exclusion of values below the LOD) to assess the robustness of the imputation strategies.

Branched isomers of PFHxS, PFHpS, PFOS, PFNS, PFDS, and PFOSA will be calculated as: Branched = sum – linear.

The difference in PFAS concentrations within each group from baseline at W1 to the end point at W18 between the study groups will be estimated using generalized linear models (or similar methods). For continuous outcomes, we will use an identity link function and assume a Gaussian distribution family.

We will also consider analyses using other distribution families based on the skewness of the data, as well as whether to categorize (e.g., dichotomize) the outcome variable.

We will also consider quantile regression and express the effects as the median differences between the study groups.

Bootstrap confidence intervals (95%) for median concentrations and median changes will be calculated using 1,000 resampling iterations to provide robust estimates that are not sensitive to non-normality.

We will also use mediation analyses to estimate the extent to which the effect is mediated through changes in albumin concentration.

### Results

### **Figures**

Flow chart of participants and samples, including ITT and PP populations and the number of donations.

Plots showing the concentration of different PFAS from week 1 to week 18.

#### **Tables**

Table 1: Baseline characteristics

| | HFPDs | RFPDs | Control group |
|----------------------------|-------|-------|---------------|
| Age | | | |
| Height | | | |
| Weight | | | |
| BMI | | | |
| Donation history | | | |
| <ul> <li>Plasma</li> </ul> | | | |
| Whole blood | | | |
| Occupation | | | |

Table 2: Baseline concentration of PFAS (incl. branched and linear isomers)

| | HFPDs | RFPDs | Control group |
|--------------|-------|-------|---------------|
| PFBA (ng/mL) | | | |
| ••• | | | |

Table 3: Concentrations of PFAS at W18 and change from W1

| PFAS | HFPDs | | RFPDs | | Control group | |
|---------|-------|------|-------|------|---------------|--------|
| | W18 | W18- | W18 | W18- | W18 | W18-W1 |
| | | W1 | | W1 | | |
| PFBA | | | | | | |
| (ng/mL) | | | | | | |
| ••• | | | | | | |

<sup>\*</sup>p-value compared to controls at W18

# Ethical considerations and data storage

All data and analyses are securely stored and managed on a safe dedicated server at Innlandet Hospital Trust. This study was funded by Innlandet Hospital Trust, Norway.

# Supplementary

Table S1: Individual limits of detection (LODi) of PFAS:

| PFAS | Range | Median | Mean |
|--------------|-------|--------|------|
| PFBA (ng/mL) | | | |

**Table S2:** Detection frequencies of analysed PFAS in all samples and per intervention group.

| PFASs | All | All | All | HFPD | | RFPD | | Control | |
|---|---|---|---|---|---|---|---|---|---|
| | samples | samples | samples | W1 | W18 | W1 | W18 | W1 | W18 |
| | | W1 | W18 | | | | | | |
| PFBA | | | | | | | | | |
| (ng/mL) | | | | | | | | | |
| ••• | | | | | | | | | |

Data are n (%)>LOD (n (%)>LOQ).

# **Authorship**

Authorship for this paper will be determined based on the Vancouver Convention on authorship [16]:

Morten Haugen (MH, corresponding and first author)

Karin Magnussen (KM)

Sandra Huber (SH)

Lise Sofie Haug Nissen-Meyer (LSHNM)

Tor A. Strand (TAS)

The order of authorship may be revised according to the authors' respective contributions.

# Timeline and Responsibilities

| Task | Deadline | Responsibility |
|---|---|---|
| Completion and approval of SAP | August 2025 | MH, SH, KM, TAS, LSHNM |
| Completion of data set | August 2025 | MH, TAS |
| Drafting introduction and methods section | August 2025 | MH, SH |

| Task | Deadline | Responsibility |
|---|---|---|
| Statistical analysis | September 2025 | MH, TAS, LSHNM |
| Drafting results section | September/October 2025 | MH, SH |
| Drafting discussion section | October 2025 | MH, SH |
| Evaluation of paper draft | November/December 2025 | MH, SH, KM, TAS, LSHNM, |
| Final manuscript submission | December 2025/January<br>2026 | МН |

### References

- Evich MG, Davis MJB, McCord JP, Acrey B, Awkerman JA, Knappe DRU, et al. Per- and polyfluoroalkyl substances in the environment. Science. 2022; 375: eabg9065.
- Buck RC, Franklin J, Berger U, Conder JM, Cousins IT, de Voogt P, et al. Perfluoroalkyl and polyfluoroalkyl substances in the environment: terminology, classification, and origins. Integr Environ Assess Manag. 2011; 7: 513–41.
- Meegoda JN, Kewalramani JA, Li B, Marsh RW. A Review of the Applications, Environmental Release, and Remediation Technologies of Per- and Polyfluoroalkyl Substances. Int J Environ Res Public Health. 2020; 17.
- Moro G, Liberi S, Vascon F, Linciano S, De Felice S, Fasolato S, et al. Investigation of the Interaction between Human Serum Albumin and Branched Short-Chain Perfluoroalkyl Compounds. Chem Res Toxicol. 2022; 35: 2049–58.
- Alesio JL, Slitt A, Bothun GD. Critical new insights into the binding of poly- and perfluoroalkyl substances (PFAS) to albumin protein. Chemosphere. 2022; 287: 131979.
- Forsthuber M, Kaiser AM, Granitzer S, Hassl I, Hengstschläger M, Stangl H, et al. Albumin is the major carrier protein for PFOS, PFOA, PFHxS, PFNA and PFDA in human plasma. Environ Int. 2020; 137: 105324.
- Lu Y, Meng L, Ma D, Cao H, Liang Y, Liu H, et al. The occurrence of PFAS in human placenta and their binding abilities to human serum albumin and organic anion transporter 4. Environ Pollut. 2021; 273: 116460.
- 8 Agency. EC. Per- and polyfluoroalkyl substances (PFAS). Available from: https://echa.europa.eu/hot-topics/perfluoroalkyl-chemicals-pfas. Last accessed 1 September 2025.
- 9 Fenton SE, Ducatman A, Boobis A, DeWitt JC, Lau C, Ng C, et al. Per- and Polyfluoroalkyl Substance Toxicity and Human Health Review: Current State of Knowledge and Strategies for Informing Future Research. Environ Toxicol Chem. 2021; 40: 606–30.
- Engelhardt JA, Plassmann MM, Weiss JM. An extended PFAS profiling of a Swedish subpopulation and mixture risk assessments using multiple approaches. Environ Int. 2025; 195: 109214.
- Gasiorowski R, Forbes MK, Silver G, Krastev Y, Hamdorf B, Lewis B, et al. Effect of Plasma and Blood Donations on Levels of Perfluoroalkyl and Polyfluoroalkyl Substances in Firefighters in Australia: A Randomized Clinical Trial. JAMA Netw Open. 2022; 5: e226257.
- Huber S, Brox J. An automated high-throughput SPE micro-elution method for perfluoroalkyl substances in human serum. Anal Bioanal Chem. 2015; 407: 3751–61.

- 13 Chain EPanel oCitF, Schrenk D, Bignami M, Bodin L, Chipman JK, del Mazo J, et al. Risk to human health related to the presence of perfluoroalkyl substances in food. EFSA Journal. 2020; 18: e06223.
- Berg V, Charles DD, Huber S, Nøst TH, Sandanger TM, Averina M, et al. Temporal changes in per and polyfluoroalkyl substances and their associations with type 2 diabetes. Scientific Reports. 2025; 15: 22026.
- Averina M, Huber S, Almås B, Brox J, Jacobsen BK, Furberg AS, et al. Early menarche and other endocrine disrupting effects of per- and polyfluoroalkyl substances (PFAS) in adolescents from Northern Norway. The Fit Futures study. Environ Res. 2024; 242: 117703.
- Uniform requirements for manuscripts submitted to biomedical journals: Writing and editing for biomedical publication. J Pharmacol Pharmacother. 2010; 1: 42–58.